CLINICAL TRIAL: NCT03019549
Title: Effect of LY3314814 on the Pharmacokinetics of Rosuvastatin in Caucasian Healthy Subjects
Brief Title: A Study of Lanabecestat (LY3314814) in Healthy Participants When Taken With Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15994; I8D-MC-AZEB (Other: Eli Lilly and Company.)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — lanabecestat; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Experimental): Period 1: 20 mg rosuvastatin administered once orally (PO)
  Interventions: Drug: Rosuvastatin
- Lanabecestat + Rosuvastatin (Experimental): Period 2: 50 mg Lanabecestat (LY3314814) administered orally (PO) Day 1 to Day 12 Rosuvastatin: 20 mg co-administered PO on Day 8
  Interventions: Drug: Lanabecestat; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Lanabecestat — Administered orally
  Other Names: LY3314814; AZD3293
  Arms: Lanabecestat + Rosuvastatin
Drug: Rosuvastatin — Administered orally

SUMMARY:
The purpose of this study is to evaluate the effect of lanabecestat on rosuvastatin. The amount of rosuvastatin in the blood will be compared, when taken alone, and then when taken with lanabecestat. The amount of lanabecestat that gets into the bloodstream will be measured. Information about any side effects that may occur will also be collected.

Participants will be on study for 21 days with a follow-up at least 7 days afterwards.

Screening will be undertaken within 45 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Women not of childbearing potential may participate and include those who are:

  * Infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as mullerian agenesis; or
  * Postmenopausal - defined as women over 50 years of age with an intact uterus who have not taken hormones or oral contraceptives within 1 year, who have had either Spontaneous cessation of menses for at least 12 consecutive months, or 6 to 12 months of spontaneous amenorrhea with follicle-stimulating hormone level greater than (>)40 milli-international units per millilitre (mIU/mL) consistent with menopause
* Caucasian and may be of Hispanic ethnicity
* Body mass index (BMI) of 19 to 32 kilogram per meter square (kg/m²), inclusive, at the time of screening

Exclusion Criteria:

- Have a clinically significant abnormal blood pressure or heart rate (supine) as determined by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2017-05-22 (Actual); Study Completion 2017-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

REFERENCES:
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15994&attachmentIdentifier=87713afe-ea99-4c11-b4da-b46306330ffb&fileName=CSP_NCT03019549.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=15994&attachmentIdentifier=b280b981-c986-4621-b8bd-ce2ab29f17e8&fileName=SAP_NCT03019549.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants completed Period 1 but did not enter Period 2 because they did not meet the genotype criteria.
Groups:
- Overall Study: All participants received: Period 1, Day 1: single, PO dose 20 mg rosuvastatin with a seven day wash-out. Period 2: Day 1-7 single, PO dose 50 mg lanabecestat (LY3314814) with a single 20 mg rosuvastatin dose coadminstered on Day 8
Period: Period 1
Arm/Group | Overall Study
Started | 42
Received 1 Dose of Study Drug | 42
Completed | 42
Not Completed | 0
Period: Washout
Arm/Group | Overall Study
Started | 42
Completed | 31
Not Completed | 11
Not completed — DId not meet genotype criteria | 11
Period: Period 2
Arm/Group | Overall Study
Started | 31
Received at Least 1 Dose of Study Drug | 29
Completed | 26
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All participants who received at least 1 dose of study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
Genotype rsl045642 (ABCB1) [Count of Participants; unit: Participants] — Results from genotype rsl045642 was used to explore polymorphisms in genes coding for certain transporters on the magnitude of the interaction between rosuvastatin and LY3314814.
  Participants
    Genotype A/A | 10
    Genotype A/G | 15
    Genotype G/G | 6
    Not performed | 11

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under The Drug Concentration Time Curve From Zero to Infinity (AUC-∞) of Rosuvastatin
Description: Pharmacokinetics (PK): Area Under The Drug Concentration Time Curve from Zero to Infinity (AUC-∞) of Rosuvastatin
Time Frame: 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 hours postdose
Population: All participants who received at least 1 dose of study drug, had evaluable PK parameters. Period 2 stand alone lanabecestat PK was not performed so only 2 arms are presented that is the data in totality.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanogram per milliliter
Groups:
- Rosuvastatin: 20 mg rosuvastatin administered PO
- Rosuvastatin + Lanabecestat (LY3314814): 20 mg rosuvastatin and 50 mg lanabescestat (LY3314814) administered in combination.
Arm/Group | Rosuvastatin | Rosuvastatin + Lanabecestat (LY3314814)
Number analyzed (Participants) | 31 | 26
hours times nanogram per milliliter | 80 (47) | 78 (56)

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Drug Concentration Time Curve During a 24-hour Dosing Interval (AUCτ) of Lanabecestat (LY3314814)
Description: Pharmacokinetics (PK): Area Under the Drug Concentration Time Curve During a 24-hour Dosing Interval (AUCτ) of Lanabecestat (LY3314814)
Time Frame: Period 2 (Day 7, 8): Predose, 0.5, 1, 2, 3, 4, 8, 12 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanograms per milliliter
Groups:
- Lanabecestat (LY3314814): 50 mg lanabecestat (LY3314814) PO once daily (QD)
- Rosuvastatin + Lanabecestat (LY3314814): 20 mg rosuvastatin and 50 mg lanabescestat (LY3314814) administered in combination PO
Arm/Group | Lanabecestat (LY3314814) | Rosuvastatin + Lanabecestat (LY3314814)
Number analyzed (Participants) | 26 | 26
hours times nanograms per milliliter | 3650 (25) | 3790 (21)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lanabecestat
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lanabecestat
Time Frame: .Period 2 (Day 7, 8): Predose, 0.5, 1, 2, 3, 4, 8, 12 hours postdose
Population: All participants who received at least 1 dose of study drug and had evaluable PK data. Period 2 stand alone lanabecestat PK was not performed so only 2 arms are presented that is the data in totality.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Lanabecestat (LY3314814) | Rosuvastatin + Lanabecestat (LY3314814)
Number analyzed (Participants) | 26 | 26
nanograms per milliliter | 369 (27) | 399 (20)

ADVERSE EVENTS:
Time Frame: Up to 5 months
Description: All participants who received at least 1 dose of study drug.
Groups:
- 20 mg Rosuvastatin: Period 1: rosuvastatin: 20 mg PO on Day 1
- 50 mg Lanabecestat (LY3314814): Period 2: Day 1-7,50 mg lanabecestat (LY3314814) PO once daily (QD)
- Lanabecestat (LY3314814) + 20 mg Rosuvastatin: Period 2: Lanabecestat (LY3314814) 50 mg PO Days 1-12 with a single dose of 20 mg rosuvastatin PO on Day 8
Arm/Group | 20 mg Rosuvastatin | 50 mg Lanabecestat (LY3314814) | Lanabecestat (LY3314814) + 20 mg Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 0/42 | 2/29 | 3/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Rosuvastatin (N=42) | 50 mg Lanabecestat (LY3314814) (N=29) | Lanabecestat (LY3314814) + 20 mg Rosuvastatin (N=26)
Surgical skin tear (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
11 participants completed Period 1 and then discontinued due to genotyping criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03019549/SAP_000.pdf
  • Study Protocol (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03019549/Prot_001.pdf